CLINICAL TRIAL: NCT05149261
Title: Coagulopathy in Acute Aortic Syndrome
Acronym: SAACAOG
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: European Georges Pompidou Hospital (Other)
Responsible Party: Principal Investigator, Diane Zlotnik, Principal Investigator, European Georges Pompidou Hospital
Other Study IDs: SAACOAG
Record Dates: First submitted 2021-11-08; First posted 2021-12-08 (Actual); Last update posted 2021-12-08 (Actual); Status verified 2021-11

CONDITIONS: Coagulopathy
Keywords: Coagulopathy; Acute aortic dissection; Blood transfusion
MeSH Terms: conditions — Hemostatic Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Routine care blood samples will be taken at different moments of the hospital stay
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Acute aortic syndrome: patients admitted to the Georges Pompidou European Hospital via the "SOS aorta" network

SUMMARY:
The existence of AAS coagulopathy has been reported, related to blood contact with the walls of the non-endothelialized false lumens. It is likely that endothelial dysfunction generated by vascular lesions may largely contribute to the development of coagulopathy, such as described in trauma-induced coagulopathy. This endotheliopathy of the AAS has never been evaluated. The coagulopathy of AAS and more specifically the endotheliopathy are poorly described and therefore have no standardized treatment.

The main objective of this study is to describe the coagulopathy

DETAILED DESCRIPTION:
Acute aortic syndromes (AAS) result from an organic lesion of the aortic wall. The various symptoms of AAS, mainly the acute chest pain, leads to a breakdown of the intima or the media of the aorta. This syndrome is made of three entities : aortic dissection (DA), intra-mural hematoma (HIM) and penetrating atherosclerotic ulcer (PAU). Surgery is a complex emergency treatment of choice. Patients suffering from these pathologies die mainly from hemorrhagic shock due to haemostasis disorders, which requires massive transfusion. The existence of AAS coagulopathy has been reported, related to blood contact with the walls of the non-endothelialized false lumens. It is likely that endothelial dysfunction generated by vascular lesions may largely contribute to the development of coagulopathy, such as described in trauma-induced coagulopathy. This endotheliopathy of the AAS has never been evaluated. The coagulopathy of AAS and more specifically the endotheliopathy are poorly described and therefore have no standardized treatment.

The main objective of this study is to describe the coagulopathy and more specifically the endotheliopathy of AAS, in particular assessing coagulation disorders, hyperactivation of fibrinolysis, quantitative or functional platelets disorder and endotheliopathy. The secondary objective is to determine the factors associated with this coagulopathy. This includes 1 / assessment of potential risk factors for coagulopathy, 2 / the prognosis of coagulopathy by assessing the relationship between coagulopathy and transfusion requirements and mortality.

ELIGIBILITY:
Inclusion Criteria:

* admitted to hospital via the "SOS Aorta" network for acute aortic syndrome (AAS) suspicion

Exclusion Criteria:

* aged < 18y
* pregnant women
* no social security

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: The EGPH offers, since 2009, a multidisciplinary network called "SOS Aorta" to centralize clinico-radiological suspicions of acute aortic syndrome in Ile de France and provide responsive and accessible medico-surgical care permanently. We included prospectively and analysed retrospectively (descripive study) all patient aged more than 18y who were admitted at EGPH for AAS suspicion via SOS Aorta Network.
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2019-07-01 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
total transfusion requirements | Day 2
  red blood cells units (number)
death from AAS | Day 30
  probability of Survival (pourcentage %)
coagulopathy rTQ > 1.2 incidence | baseline
  pourcentage %

SECONDARY OUTCOMES:
total transfusion requirements | Day 1
  red blood cell unit, fresh frozen plasma and platelets units (number)
total transfusion requirements | Day 2
  red blood cell unit, fresh frozen plasma and platelets units (number)
total transfusion requirements | Day 3
  red blood cell unit, fresh frozen plasma and platelets units
total transfusion requirements | Day 7
  red blood cell unit, fresh frozen plasma and platelets units
biological AAS coagulopathy : coagulation factors consumption | Day 1, Day 2, Day 3, Day 7
  pourcentage %
biological AAS coagulopathy : coagulation factors consumption | Day 2
  pourcentage %
biological AAS coagulopathy : coagulation factors consumption | Day 3
  pourcentage %
biological AAS coagulopathy : coagulation factors consumption | Day 7
  pourcentage %
biological AAS coagulopathy : fibrinolysis D-dimers | Day 1
  µg/L
biological AAS coagulopathy : fibrinolysis D-dimers | Day 2
  µg/L
biological AAS coagulopathy : fibrinolysis D-dimers | Day 3
  µg/L
biological AAS coagulopathy : fibrinolysis D-dimers | Day 7
  µg/L
hospitalisation duration | hospital discharge
  number of days
impact of misdiagnosis and misdiagnosis-induced treatments | Day 2
  massive post-operative bleeding (BART definition)
impact of misdiagnosis and misdiagnosis-induced treatments | Day 7
  massive post-operative bleeding (BART definition)
platelets dysfunction | day 1
  platelets rate G/L
platelets dysfunction | day 2
  platelets rate G/L
platelets dysfunction | day 3
  platelets rate G/L
platelets dysfunction | day 7
  platelets rate G/L
platelets dysfunction | baseline
  CD 40 L pg/mL
endotheliopathy | baseline
  IL6 rate pg/mL
endotheliopathy | baseline
  IL8 rate pg/mL
endotheliopathy | baseline
  syndecan rate pg/mL
endotheliopathy | baseline
  endocan rate pg/mL
endotheliopathy | baseline
  angiopoietine 2 rate ng/mL
endotheliopathy | baseline
  angiopoietine 2 / angiopoietine 2 ratio
endotheliopathy | baseline
  VEGF ng/mL
endotheliopathy | baseline
  FGF basic ng/mL
symptoms-surgery delay | baseline
  time hours
clinical severity shock | baseline
  acidosis pH
clinical severity shock | baseline
  lactate level (mmol/L)
clinical severity shock | baseline
  number of organs with malperfusion (number)

CONTACTS AND LOCATIONS:
Overall Officials: Diane Zlotnik, MD, Principal Investigator — European Georges Pompidou Hospital; Anne Godier, MD-PhD, Study Chair — European Georges Pompidou Hospital
Locations (1):
- Université de Paris, Paris, France

IPD SHARING:
Plan to Share IPD: Undecided
we will maybe try later to make a multicentric descriptive analysis with other french hospitals